CLINICAL TRIAL: NCT07113613
Title: A Multicenter, Single-arm Phase II Clinical Study on Exempting Tumor Bed Boost Radiotherapy for Patients Achieving pCR After Breast Conserving Surgery With Neoadjuvant Therapy
Brief Title: Prospective Study on Exemption of Tumor Bed Boost Radiotherapy for pCR Patients After Breast Conserving Surgery With Neoadjuvant Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Sun Xinchen, Director of the Radiotherapy Center, The First Affiliated Hospital with Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-SR-983
Record Dates: First submitted 2025-08-06; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
Keywords: Radiotherapy; Exemption of tumor bed dosage increase; Breast-conserving treatment; Neoadjuvant chemotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exempted tumor bed radiotherapy group (Experimental): The total breast irradiation dose was 43.5 Gy/15 fractions, with each fraction being 2.9 Gy, administered once a day, 5 times a week; the dose for the regional lymph nodes was also 43.5 Gy/15 fractions, with each fraction being 2.9 Gy, administered once a day, 5 times a week.
  Interventions: Radiation: Exemption from additional radiotherapy on the tumor bed after surgery

INTERVENTIONS:
Radiation: Exemption from additional radiotherapy on the tumor bed after surgery — For patients who met the inclusion criteria and were enrolled, postoperative tumor bed boost radiotherapy was waived, and only whole breast and/or regional lymph node irradiation was administered.

SUMMARY:
This study is a multicenter, single-arm, phase II clinical trial, aiming to evaluate the safety and efficacy of tumor bed dose escalation radiotherapy for patients with primary breast lesions achieving pCR (ypT0) after neoadjuvant chemotherapy and breast-conserving surgery.

DETAILED DESCRIPTION:
New neoadjuvant chemotherapy (NAC) is mainly used for patients with locally advanced or those who wish to preserve their breast. It not only helps to downstage the tumor but also increases the success rate and possibility of breast-conserving treatment for patients. Moreover, NAC provides doctors with the opportunity to assess the chemotherapy response, which can be used to predict the survival of patients. Studies have shown that patients who achieve pathological complete response (PCR) after NAC and surgery have a lower local-regional recurrence rate, higher disease-free survival rate and overall survival rate. Currently, there are no treatment guidelines for this group of patients. Avoiding unnecessary tumor bed dose escalation can reduce radiotherapy toxicity and help promote the effective utilization of medical resources. This study is the first prospective single-arm study to explore the prognostic significance of NAC and breast-conserving surgery without tumor bed dose escalation for patients with pCR breast cancer. The aim is to identify the appropriate population for exemption from tumor bed dose escalation and to develop more precise adjuvant radiotherapy plans.

ELIGIBILITY:
Inclusion Criteria:

(1) Voluntary participation, good compliance, able to cooperate with the trial observation, and having signed a written informed consent form; (2) Confirmed as invasive cancer through pathological tissue examination, and received baseline breast MR or PET/MR examination before neoadjuvant therapy; (3) Received the standard neoadjuvant treatment plan recommended by the guidelines based on molecular typing; (4) Single lesion, initially diagnosed as cT1-3N0-3a; (5) Underwent breast-conserving surgery, with negative surgical margins and a margin distance of ≥1mm, and achieved pCR of the primary breast lesion after NAC (ypT0); (6) Age 30-75 years, ECOG score 0-1; (7) Met the basic requirements for adjuvant radiotherapy, including basically normal peripheral blood count, no significant abnormalities in heart, liver, and kidney functions, and basically normal electrocardiogram; (8) Had no previous chest radiotherapy.

Exclusion Criteria:

(1) Pregnant women, lactating women, or women with reproductive capacity but without contraceptive measures in place; (2) Known to carry mutated susceptibility genes for breast cancer (including BRCA-1 and BRCA-2); (3) Diagnosed with cT4, N3b-c, bilateral breast cancer, with multiple primary lesions, multicentricity or non-bulky enhancement at the primary site; (4) Not receiving the standard neoadjuvant treatment regimen recommended by guidelines, or the primary breast lesion did not achieve pCR (including ypTis) after NAC; (5) Suffering from other malignant tumors or participating in other clinical trials simultaneously; (6) Unable to start radiotherapy within 8 weeks after breast cancer surgery; (7) Diagnosed with distant metastasis through initial imaging or pathology; (8) Previous history of breast cancer, history of radiotherapy in the neck, chest or ipsilateral axilla; (9) Severe non-tumor-related medical comorbidities affecting the implementation of radiotherapy; (10) Suffering from uncontrollable neurological, mental disorders or mental impairments, with poor compliance and inability to cooperate and describe treatment responses.

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study only included female breast cancer patients.
Enrollment: 150 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
5-year ipsilateral breast recurrence rate (IBTR) | 5 years
  The recurrence of the same-sided breast occurred for the first time within 5 years.
5-year local-regional recurrence (LRR) | 5 years
  Recurrence of the same-side breast, the same-side axillary fossa, the same-side supraclavicular lymph nodes, or the same-side internal mammary lymph nodes for the first time within 5 years.

SECONDARY OUTCOMES:
Local regional control rate (LRC) | 5 years
  The time from NAC to the occurrence of the first LRR
Disease-free survival time (DFS) | 5 years
  The time from NAC to recurrence or death
Overall survival time (OS) | 5 years
  The time from chemotherapy to death due to any cause
Safety-related study endpoints | 5 years
  acute or chronic radiotherapy-related adverse reactions: including skin damage, breast pain, lung damage, heart damage, upper limb edema, upper limb functional impairment, brachial plexus injury, etc.
cosmetic effect | 5 years
  evaluation of cosmetic effect after breast-conserving surgery using the Harvard standard.
quality of life evaluation | 5 years
  quality of life evaluation using the Chinese version of the QLQ-BR23 scale.

CONTACTS AND LOCATIONS:
Overall Officials: Xinchen Sun, Doctor, Principal Investigator — The First Affiliated with Nanjing Medical University (Jiangsu Province People's Hospital)
Locations (1):
- The First Affiliated with Nanjing Medical University (Jiangsu Province People's Hospital), Nanjing, Jiangsu, China